CLINICAL TRIAL: NCT01369524
Title: Evaluation of Effect of Fluid Resuscitation on Sublingual Microcirculation by SDF Imaging in Intensive Care Patients, a Pilot Study
Brief Title: Effect of Fluid Resuscitation and Microcirculation
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Dr E.C. Boerma, Medical Centre Leeuwarden
Other Study IDs: TPO 732
Record Dates: First submitted 2011-05-31; First posted 2011-06-09 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-05

CONDITIONS: Total Fluid Volume Increased
Keywords: fluid responsiveness; microcirculation; Intensive Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICUpatient with need of fluid: age > 18 - haemodynamic monitoring - informed consent - admission on ICU

SUMMARY:
Although the investigators take many measurements to monitor the fluid state of the patients, it is not known exactly whether the fluid has real effect on the organ perfusion. The main focus of fluid is to improve the organ perfusion. Recent research has focused on the investigation of sublingual microcirculatory alterations.

DETAILED DESCRIPTION:
Is fluid responsiveness, what means a better cardiac output, equal to the need for fluid for a better organ perfusion? In hospital the investigators are now looking to the pump function of the heart, as there is not a better measurement. However this gives no information about necessity of giving fluids. A healthy volunteer also gives a better pump function of the heart after fluid, but that fluid is not necessary and gives no better organ perfusion. The question is: How many percent of the patients have a MFI score of < 2.6, when the doctor on clinical basis plans to give fluid to the patient, improves organ perfusion after fluid, and is this correlated with an improvement of the cardiac output All intensive care patients who need extra fluid are eligible for this study. Before and after the fluid challenge we do SDF imaging sublingual. Per patient the investigators do this 1x in 24 hours. Concurrently, data on both patient characteristics (e.g. severity of illness) will be obtained Study population max 100 patients. Possible outcome: MFI < 2,6 en SV > 10% + MFI up MFI < 2,6 en SV equal + MFI equal MFI < 2,6 en SV > 10% + MFI equal MFI < 2,6 en SV equal + MFI up MFI > 2,6 en SV > 10% + MFI up MFI > 2,6 en SV equal + MFI equal MFI > 2,6 en SV > 10% + MFI equal MFI > 2,6 en SV equal + MFI up

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* hemodynamic monitoring
* informed consent
* admission on ICU

Exclusion Criteria:

* no informed consent
* oral surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted on the ICU and a need of fluids
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
correlation between change in microvascular flow index and fluid responsiveness - delta MFI before and after fluid challenge correlated to fluid responsiveness | 24 hours

SECONDARY OUTCOMES:
change in capillary density correlated to fluid responsiveness | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Boerma, MD, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Medical Centre Leeuwarden, Leeuwarden, Netherlands